CLINICAL TRIAL: NCT02927626
Title: Clinical Research of Yang Yin Fu Zheng Therapy in HBV Associated Hepatocellular Carcinoma Basing on Immune Microenviroment
Brief Title: Yang Yin Fu Zheng Therapy in HBV Associated Hepatocellular Carcinoma
Acronym: YYFZTIHBVHCC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Zhiyun Yang, archiater,professor, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingDH
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

ARMS (2):
- Yang Yin Fu Zheng therapy (Experimental)
  Interventions: Drug: Yang Yin Fu Zheng therapy; Drug: Routine medical care
- Routine medical care (Placebo Comparator)
  Interventions: Drug: Routine medical care

INTERVENTIONS:
Drug: Yang Yin Fu Zheng therapy — Yang Yin Fu Zheng is a Chinese herbal compound.
  Arms: Yang Yin Fu Zheng therapy
Drug: Routine medical care — Routine medical care

SUMMARY:
Clinical research of Yang Yin Fu Zheng therapy in HBV associated hepatocellular carcinoma basing on immune microenviroment.The purpose of this study is to observe the efficacy of routine medical care combined with Yang Yin Fu Zheng therapy for patients belong to HBV-HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed of stage HBV-HCCⅡb、Ⅲa、Ⅲb;
2. Ages Eligible for Study: ≤75 years old;
3. TCM syndrome is deficiency of both Qi and Yin;
4. Confirmed of CHB;
5. Surgery cannot be allowed;
6. Informed consent from the patient.

Exclusion Criteria:

1. Patient with other chronic hepatopathy, such as AIH, NAFLD, ALD;
2. Serious problem of heart, lung, or kidney with severe dysfunction;
3. Pregnant or child breast feeding women;
4. Mental or cognitive disorders;
5. Participating in other drug trials;
6. Who are allergic to the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Survival rate | 2 years

SECONDARY OUTCOMES:
Objective response rate | 2 years
quality of life(QOL) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyun Yang, PhD, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Zhiyun Yang, Beijing, Beijing Municipality, China